CLINICAL TRIAL: NCT05040789
Title: A Randomized, Observer-Blind, Multicenter, Phase 3 Study to Evaluate the Lot Consistency of a Recombinant Coronavirus-Like Particle COVID-19 Vaccine in Adults 18-49 Years of Age
Brief Title: Phase 3 Study to Evaluate the Lot Consistency of a Recombinant Coronavirus-Like Particle COVID-19 Vaccine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Further development terminated
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-PRO-CoVLP-024
Record Dates: First submitted 2021-08-26; First posted 2021-09-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): CoVLP Lot 1
  Interventions: Biological: CoVLP formulation
- Group 2 (Experimental): CoVLP Lot 2
  Interventions: Biological: CoVLP formulation
- Group 3 (Experimental): CoVLP Lot 3
  Interventions: Biological: CoVLP formulation

INTERVENTIONS:
Biological: CoVLP formulation — The Coronavirus-Like Particle (CoVLP) COVID-19 Vaccine is composed of recombinant spike (S) glycoprotein expressed as virus-like particles (VLPs).
  The 3.75 µg dose of CoVLP will be administered with the adjuvant AS03 (manufactured by GlaxoSmithKline).

SUMMARY:
This Phase 3 study is intended to assess clinical lot-to-lot consistency by evaluating and comparing the immunogenicity of three consecutively manufactured lots of Coronavirus-like Particle (CoVLP).

DETAILED DESCRIPTION:
This is a randomized, observer-blinded, multicenter, Phase 3 lot-to-lot consistency study in approximately 900 healthy seronegative adults 18-49 years of age after the administration of two doses of CoVLP (3.75 ug) adjuvanted with AS03 (referred to as "CoVLP formulation").

Subjects who are seronegative for SARS-CoV-2 antibodies will be randomized in a 1:1:1 ratio to receive one of three lots of the CoVLP formulation. Subjects will receive two intramuscular injections 21 days apart. The same lot will be used for both IM injections in each subject. Safety and immunogenicity assessments will be performed. Subjects will participate in this study for approximately 49 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be 18 - 49 years of age at screening visit.
* Subjects must have a body mass index < 35 kg/m2 at screening visit.
* Subjects must be in good general health prior to study participation. Note: Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and the condition is unlikely to confound the results of the study or pose additional risk to the subject.
* Female subjects of childbearing potential must have a negative urine pregnancy test result prior to vaccination.
* Female subjects of childbearing potential must use a highly effective method of contraception starting one month prior to vaccination, continuing until the end of the study, and must not plan to become pregnant for at least one month after her last study vaccination.

Exclusion Criteria:

* Significant acute or chronic, uncontrolled medical or neuropsychiatric illness.
* Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, human immunodeficiency virus (HIV), hepatitis B or C infection (subjects with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time are allowed).
* Current autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus or multiple sclerosis).
* Administration of any medication or treatment that may alter the vaccine immune responses, such as:

  * Systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for 10 or more days in total, within one month prior to the Vaccination visit (Visit 2). Inhaled, nasal, ophthalmic, dermatological, and other topical glucocorticoids are permitted.
  * Cytotoxic, antineoplastic, or immunosuppressant drugs - within 36 months prior to Vaccination (Visit 2).
  * Any immunoglobulin preparations or blood products, blood transfusion - within 6 months prior to Vaccination (Visit 2).
* Administration of any vaccine within 14 days prior to Vaccination (Visit 2); planned administration of any vaccine during the study (up to Day 28 of the study).
* Administration of any other SARS-CoV-2 / COVID-19, or other experimental coronavirus vaccine at any time prior to or during the study.
* History of virologically-confirmed COVID-19.
* Use of any investigational or non-registered product within 30 days or 5 half-lives, whichever is longer, prior to Vaccination (Visit 2) or planned use during the study period.
* Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site that may interfere with injection site reaction rating.
* Use of any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that are thought to be effective for prevention of COVID-19 but have not been licensed for this indication, within one month prior to Vaccination (Visit 2).
* History of a serious allergic response to any of the constituents of CoVLP including AS03.
* History of a documented anaphylactic reactions to plants or plant components (including tobacco, fruits and nuts).
* Personal or family (first-degree relatives) history of narcolepsy.
* Subjects with a history of Guillain-Barré Syndrome.
* Any female subject who has a positive or doubtful pregnancy test result prior to vaccination or who is lactating.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-22 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
GMTs of the three vaccine lots | Up to Day 42 (21 days after the second vaccination)
  Nab response induced against the SARS-CoV-2 virus on Day 42 will be analyzed using GMTs of the three vaccine lots on Day 42 adjusted for Day 0 GMTs.

SECONDARY OUTCOMES:
Immediate adverse events | 30 minutes after each vaccine administration
  Occurrence, intensity, and relationship to vaccination of immediate adverse events.
Solicited adverse events | Seven days following each vaccination
  Occurrence and intensity of solicited local and systemic adverse events.
Unsolicited adverse events | 21 days following each vaccination
  Occurrence, intensity, and relationship of unsolicited adverse events.
Other adverse events | Up to 21 days following each vaccine administration
  Occurrences of serious AEs (SAEs), medically attended AEs (MAAEs), AEs leading to withdrawal, AE of special interest (AESIs; including vaccine-associated enhanced disease [VAED], anaphylaxis, and severe allergic reactions), and deaths.
SC rates | 21 days after the second vaccination
  Nab response induced by CoVLP (3.75 µg/dose) adjuvanted with AS03 against the SARS-CoV-2 virus on Day 0 and Day 42 will be analyzed using SC rates
GMFRs | 21 days after the second vaccination
  Nab response induced by CoVLP (3.75 µg/dose) adjuvanted with AS03 against the SARS-CoV-2 virus on Day 0 and Day 42 will be analyzed using GMFRs

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dawson Clinical Research, Guelph, Ontario
  - LMC Manna Research, Toronto, Ontario